CLINICAL TRIAL: NCT03326934
Title: The Impact of Chocolate on Visual Performance: Psychophysics and Electrophysiology
Brief Title: Impact of Dark Chocolate on Visual Performance
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of the Incarnate Word (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Basic Science
Other Study IDs: 17-06-002
Record Dates: First submitted 2017-10-19; First posted 2017-10-31 (Actual); Last update posted 2019-04-18 (Actual); Status verified 2019-04

CONDITIONS: Dietary Supplementation

STUDY DESIGN:
Intervention Model Description: Randomized, single-masked crossover study to assess potential effects of dark chocolate vs. milk chocolate on multiple aspects of visual function and performance.
Who Masked: Participant
Masking Description: None of the subjects will be aware of the intent of the study to the type of chocolate consumed prior to each of two testing sessions
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Milk Chocolate (Sham Comparator): Each subject consumes a Trader Joe's Crispy Rice Milk Chocolate bar: 40g, 12.4g milk chocolate cocoa; total flavanols: 40 mg.
  Interventions: Dietary Supplement: Milk Chocolate
- Dark Chocolate (Experimental): Each subject consumes a Trader Joe's 72% Cacao Dark Chocolate bar: 47g, 34g cacao, total flavanols: 316.3 mg.
  Interventions: Dietary Supplement: Dark chocolate

INTERVENTIONS:
Dietary Supplement: Dark chocolate — Trader Joe's 72% Cacao Dark Chocolate bar, 47g, 34g cacao, total flavanols: 316.3 mg.
  Arms: Dark Chocolate
Dietary Supplement: Milk Chocolate — Trader Joe's Crispy Rice Milk Chocolate bar: 40g, 12.4g milk chocolate cocoa; total flavanols: 40 mg.
  Arms: Milk Chocolate

SUMMARY:
The purpose is to conduct a randomized, single-masked crossover study to determine if acute consumption of a commercially available, highly palatable dark chocolate bar can improve visual performance. Vision testing will include multiple measures of contrast and color perception, reaction time, effects of distraction on visual performance during simulated hands-free phone calls, simulated marksmanship, as well as multiple, objective electro-diagnostic tests including standard and color visual-evoked potentials and various types of electro-retinograms to assess visual pathway function.

DETAILED DESCRIPTION:
Consumption of dark chocolate has been associated with improved blood flow, cardiovascular function, slowing of degenerative aging processes, as well as enhanced mood and cognitive performance. Dark chocolate is rich in cocoa flavanols which have both antioxidant effects to prevent and impede degenerative disease and as well as more immediate effects on local and cerebral blood flow. One study demonstrated an improvement in contrast sensitivity (CS) which is the visual ability to detect low contrast targets. Hence dark chocolate may enhance vision during critical task performance in military and law enforcement settings as well as every-day tasks such as driving. Whereas it is assumed that visual enhancements from dark chocolate derive from increased cerebral and/or retinal blood flow, direct measurements are lacking. Prior research demonstrated that hands free phone communication (verbal distraction) can delay reaction time and impair CS. Hence in this study our purpose is to determine if acute consumption of dark chocolate impacts: CS and reaction time with and without verbal distraction, measures of high and low contrast vision as well as color vision, and bjective electrophysiological measures of retinal, optic nerve and cortical function. In prior studies of acute effects of dark chocolate on cognition and CS, the dark chocolate was consumed 90-120 minutes prior to testing. In this study the investigators are using a somewhat larger dose and beginning electrophysiological testing after consumption with color and CS testing approximately 1 hour and 30 minutes afterconsumption. The investigators believe this will capture possible more immediate blood flow changes in retina and cortex based on electrophysiological measures and CS and cognitive changes later in the session.

A total of 30 subjects will be recruited from UIW and RSO students, staff, faculty and patients. The age range will be 18 to 65 years and the investigators will attempt to include comparable numbers of male and female participants. Inclusion criteria include visual acuity of at least 20/20 in each eye with no evidence of ocular, systemic or neurologic disease or ocular trauma. Based on prior research using repeated-measures designs, a difference of 0.1 log CS is considered significant and the estimated standard deviation is 0.13 log units. Hence the effect size = (mean difference)/SD = 0.1/0.13 = 0.76. The estimated minimum number of subjects to achieve significance at the 5% level with a power of 80%: (1/effect size)2 x 16 = (1/0.76)2 x 16 = 28 subjects.(8,9). Hence 30 subjects will be recruited to account for subject attrition during the course of the study. Prior to obtaining written informed consent, each subject will be briefed on the nature of the study by one or more members of the research team. Subjects will be informed that they will be evaluated with standard vision tests one hour after consuming a chocolate bar to assess its effects on performance. The dark chocolate and milk chocolate bars to be used are commercially available from Trader Joe's and have comparable ingredients and nutrients except for the higher percentage (72%) of cacao dark chocolate in the experimental bar while the control bar contains 31% milk chocolate cocao solids which are not associated with acute beneficial effects on performance. As stated in the informed consent document, subjects will be asked if they have allergies to any of the ingredients contained in the chocolate bars, and will be excluded from participating if they answer affirmatively. As noted above, any subjects with ocular, systemic or neurologic disease, including diabetes and hypoglycemia, will not be allowed to participate in the study.

A single-blinded crossover design will be used to assess possible effects of the dark or milk chocolate bars (72% cacao dark chocolate) on visual performance and visual electrophysiological signals. Double-blinding (experimenter unaware of the type of chocolate) is not tenable due to the difference in coloration and aroma of the two chocolate bars and not likely to be a significant source of variability given the objective nature of the visual performance measures. Subjects will be tested in two one-hour sessions separated by at least 72 hours. Each subject will consume a different chocolate bar one-hour prior to testing with the order of bars (dark vs. milk chocolate) counter-balanced across subjects. Subjects will be asked to refrain from consuming coffee or caffeinated drinks on the day of testing and to consume the bar without milk or milk products which can lessen beneficial effects of dark chocolate. The subject will be presented the bar in its original wrapper but with the name masked by tape and she/he will be given a paper plate and napkins and asked to remove and return the wrapping to the research team member(s). The subject will be offered water during consumption of the bar which will take place in the research room. Insofar as many of the subjects will be in-house student volunteers, she/he will then remain in UIWRSO to study, work-study, finish clinical records, etc. for about 30 minutes. The patient will then undergo preliminary evaluation to prepare for the testing to commence at least 1 hour after chocolate bar consumption. This will include measurement of distant visual acuity followed by refraction to best visual acuity if the patient does not achieve 20/20 in each eye with their habitual correction. Hence the patient will either wear their habitual correction or lenses in a trial frame to achieve best vision during testing. The patient will then be prepped for electro-diagnostic testing including visual-evoked potentials (VEPs) and electro-retinograms (ERGs) which objectively assess visual cortical and retina/optic nerve function, respectively. VEPs will be recorded using the Diopsys® system. The subject is seated comfortably before a reversing checkerboard display. The back of the head, forehead and temple will be wiped clean using an FDA approved non-abrasive cleaner. High and low contrast VEPs will be recorded from the back of the head using disposable skin electrodes with reference and ground electrodes at the forehead and temple, respectively. Cone specific color VEPs10 will also be recorded using the Diagnosys, LLC system. All VEPs will be recorded binocularly and not be initiated until one-hour following consumption of the chocolate bar. The Diopsys® system will be used to record pattern ERGs (optic nerve function), flicker ERGs (cone function) and the photopic negative response (phNR; cone, bipolar cell and optic nerve function). Half of the subjects in control and experimental sessions will be tested with ERGs first and half with VEPs first to control for order effects. These FDA approved electro-diagnostic tests will be followed by letter chart measures of large and small CS (Precision Vision, Inc.). Each subject will then be tested with the Innova Systems, Inc. computer controlled Cone Contrast Test which assesses red, green and blue cone CS as well as large and small black/white letter CS using an adaptive staircase (like a hearing test) to determine the lowest visible contrast and overall response time. As described in our previous study,7 each subject will undergo computer-based CS testing with and without verbal distraction during testing with order counterbalanced across subjects. The verbal distraction will be broadcast on a hands-free blue-tooth device to simulate an incoming phone call consisting of scripted questions to assess memory and cognitive performance while completing the CS tasks. Following these tests, the subject will be asked to perform a brief (<10 minute) Wii™ shooting game using the Wii™ zapper which is shaped like a small rifle-no training is necessary. Two-way repeated measures ANOVA will be used to assess CS across distraction and chocolate bar conditions and post-hoc paired t-tests conducted to identify specific differences. Within subject ANOVAs and post-hoc t-test comparisons also will be used to assess amplitude and latency parameters of VEPs and ERGs across dark and milk chocolate conditions.

ELIGIBILITY:
Inclusion Criteria:

* Visual acuity of at least 20/20 in each eye
* Absence of ocular disease
* Absence of ocular trauma
* Absence of systemic disease
* Absence of neurologic disease

Exclusion Criteria:

* Visual acuity less than 20/20 in either eye
* Presence of ocular disease
* Presence or history of ocular trauma
* Presence of systemic disease
* Presence of neurologic disease

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 57 (Actual)
Dates: Start 2017-06-25 (Actual); Primary Completion 2018-08-30 (Actual); Study Completion 2018-08-30 (Actual)

PRIMARY OUTCOMES:
Visual acuity, contrast sensitivity and color vision. | 20 minutes per session
  High and low contrast visual acuity, contrast sensitivity and color vision will be assessed using letter charts and computer generated stimuli. Thresholds will be compared using within subject repeated measures ANOVA and post-hoc paired t-tests across Dark and Milk chocolate. Z-scores may be used to combine data with different dependent variables.
Effects of distraction on visual performance during simulated hands-free phone calls. | 20 minutes per session.
  Measures of color vision contrast sensitivity and low contrast visual acuity will be measured with and without a simulated hands-free phone call. will be compared using within subject repeated measures ANOVA and post-hoc paired t-tests across Dark and Milk chocolate. Z-scores may be used to combine data with different dependent variables.
Visual-electrodiagnostic testing. | 60 minutes per session
  The amplitude and latency of visual brain-waves (VEPs) and eye-waves (ERGs) will be compared using within subject repeated measures ANOVA and post-hoc paired t-tests across Dark and Milk chocolate. Z-scores may be used to combine data with different dependent variables.
Simulated marksmanship. | 20 minutes per session
  A Nintendo Wii shooting game will be used to obtain accuracy scores and time for completion. Data will be expressed as throughput: ration of accuracy/time for completion. Throughput will be compared using within subject repeated measures ANOVA and post-hoc paired t-tests across Dark and Milk chocolate.

CONTACTS AND LOCATIONS:
Overall Officials: Jeff C Rabin, OD, MS, PhD, Principal Investigator — University of the Incarnate Word
Locations (1):
- University of the Incarnate Word Rosenberg School of Optometry, San Antonio, Texas, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Rabin JC, Karunathilake N, Patrizi K. Effects of Milk vs Dark Chocolate Consumption on Visual Acuity and Contrast Sensitivity Within 2 Hours: A Randomized Clinical Trial. JAMA Ophthalmol. 2018 Jun 1;136(6):678-681. doi: 10.1001/jamaophthalmol.2018.0978. PMID 29710322

DOCUMENTS (2):
  • Informed Consent Form (2018-06-20): https://cdn.clinicaltrials.gov/large-docs/34/NCT03326934/ICF_000.pdf
  • Study Protocol (2018-06-20): https://cdn.clinicaltrials.gov/large-docs/34/NCT03326934/Prot_001.pdf